CLINICAL TRIAL: NCT00636597
Title: Prospective Evaluation of Same Day Bidirectional Endoscopy for Occult Bleeding
Brief Title: A Prospective Evaluation of Same Day Bidirectional Endoscopy for Occult Bleeding
Status: Terminated | Type: Observational
Why Stopped: Not able to find enough eligible patients (200) in last 4 years.
Sponsor: US Department of Veterans Affairs (U.S. Federal Agency)
Responsible Party: Sponsor
Organization: VA Office of Research and Development (U.S. Federal Agency)
Other Study IDs: Buff VAMC 001; 00556 (Other: VA Western NY Healthcare System, Buffalo)
Record Dates: First submitted 2008-03-07; First posted 2008-03-14 (Estimated); Last update posted 2011-10-20 (Estimated); Status verified 2011-10

CONDITIONS: Occult GI Bleeding

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 1

SUMMARY:
This study is a prospective evaluation of patients with occult (hidden) GI bleeding without iron deficiency. Such patients usually undergo a diagnostic colonoscopy as a standard of care. The study is aimed to determine any UGI-source of occult bleeding and to correlate UGI symptoms with findings. Therefore, EGD is being offered to such patients as part of research. We proposed to enroll 200 consecutive patients referred to our GI-unit for expedited diagnostic colonoscopy for positive FOBT.

DETAILED DESCRIPTION:
Occult gastrointestinal bleeding is defined as iron deficiency or fecal occult blood test (FOBT) positivity with or without anemia. Colonoscopy can detect significant pathology such as colon cancer, significant precancerous polyps, or angiodysplasia. EGD can detect pathology such as esophageal or gastric cancer, peptic ulcer disease, or vascular lesions. Here at the VA, uncomplicated referrals for occult bleeding with anemia are directly schedule for EGD and colonoscopy on the same day without prior clinic visit. Cases of FOBT positivity without anemia or upper GI symptoms usually receive only colonoscopy. Both procedures are standard of care for occult bleeding and have well established safety. The diagnostic yield of bidirectional endoscopy for occult bleeding has previously been studied with mixed results due to the variability in study design, inclusion/exclusion criteria, etc. It is unclear if presentation (iron deficiency vs fobt positivity), severity (level of iron deficiency, hct, transfusion needed), medical history (renal failure, need for Aspirin or NSAIDs etc), or symptoms (upper vs lower GI) are predictive of endoscopic findings. Of particular uncertainty is the utility of upper endoscopy in patients with isolated FOBT positivity (no iron deficiency, anemia, or upper GI symptoms). In a large retrospective study of asymptomatic patients who underwent EGD following a negative colonoscopy performed for FOBT positivity without iron deficiency (with or without anemia) showed that anemia was predictive of significant positive findings (29% vs. 8%). In a prospective study, patients with FOBT positivity without iron deficiency had same bidirectional endoscopy performed. Significant upper gi lesions were more prevalent than colonic lesions (28.6% vs. 21.8%) with a low sensitivity for predicting findings based on symptoms.

Our primary purpose is to determine if anemia or upper GI symptoms can accurately predict the presence of significant upper GI findings in patients with fobt positivity and a non-diagnostic colonoscopy. We will use this information to justify or change our current endoscopic approach to such patients.

Methods:

Study size: 200 consecutive patients

Inclusion criteria:

Outpatients referred for occult bleeding (iron deficiency or fobt positivity)

Exclusion criteria:

Overt bleeding (melena, hematochezia) Abnormal luminal imaging Prior EGD or colonoscopy within 1 year

Study flow:

1. Review all outpatient referrals for occult bleeding (iron def, fobt positive).
2. All potential patients will be contacted by phone and their enrollment/participation will be discussed. If interested we will proceed.
3. We will confirm/obtain fobtx3, full iron panel (iron, tibc, ferritin), cell count (including mcv), coags, and creatinine within 1 month of procedure (if not already done within that time).
4. We will complete a standard questionnaire as outlined below. Date will come from direct questioning and review of CPRS. This will be done by phone. Questioning will take about 15 minutes. See attached.
5. Once labs and questionnaire are obtained, pts will then be scheduled for same day colon/egd (with duodenal biopsy regardless of appearance) within 30 days performed by Dr Baichi or Dr Mehboob. Colonoscopy will be performed first. Egd will be cancelled only if colon has obvious malignancy. Other positive findings will not eliminate need for egd.
6. Patient study involvement ends after completion of procedures

Results/analysis:

EGD and colonoscopy findings will be recorded and lesions will be categorized as potential bleeding source (PBS) based on criteria outlined by others.

The data will be analyzed for diagnostic yield and statistical tests will be applied as needed to assess for predictors of positive findings.

ELIGIBILITY:
Inclusion Criteria:

* Outpatients referred for occult bleeding (iron deficiency or FOBT positivity)

Exclusion Criteria:

* Overt bleeding (melena, hematochezia)
* Abnormal luminal imaging
* Prior EGD or colonoscopy within 1 year

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Outpatients referred for GI consult due to occult bleeding (iron deficiency or FOBT positivity)
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2007-04; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
to determine if anemia or upper gi symptoms can accurately predict the presence of significant upper gi findings in patients with fobt positivity and a non-diagnostic colonoscopy. | Baseline

CONTACTS AND LOCATIONS:
Overall Officials: Shahid Mehboob, MD, Principal Investigator — VA Western New York Healthcare System at Buffalo
Locations (1):
- VA Western New York Healthcare System at Buffalo, Buffalo, New York, United States